CLINICAL TRIAL: NCT01548846
Title: Impact of Tomotherapy on Xerostomia and Quality of Life of Patients With Cancer of the Upper Aero-digestive Tract
Acronym: TOQUAL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of recrutment
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: TOQUAL
Record Dates: First submitted 2012-03-06; First posted 2012-03-08 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Head and Neck Cancer; Radiotherapy by Tomotherapy Exclusive; With or Without Concurrent Chemotherapy
Keywords: tomotherapy; xerostomy; head and neck squamous cell carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Tomotherapy — Patients receive radiotherapy by Tomotherapy for 7 weeks at the ENT

SUMMARY:
This is a study whose main objective is to evaluate prospectively the proportion of patients with severe xerostomia one year after treatment with tomotherapy for head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient (e) old (e) over 18 years
* Patients with squamous cell carcinoma of head and neck (oral cavity, oropharynx, lymphadenopathy without gateway) histologically proven.
* Patient targeted for head and neck radiotherapy by Tomotherapy exclusive with or without concurrent chemotherapy (containing platinum)
* Indication of head and neck radiotherapy bilateral
* All of the TNM stage except metastatic
* Patient has signed informed consent for participation in the study
* Mastery of the French language

Exclusion Criteria:

* History of head and neck radiotherapy
* Indication of head and neck radiotherapy unilateral
* Personal history of malignant tumors uncontrolled over the past 5 years
* History of oral sicca syndrome
* Surgical removal of one or more salivary glands (parotid, submandibular gland, sublingual gland)
* Concomitant treatment with amifostine
* Concomitant treatment with cetuximab
* Primary tumor of the salivary glands
* Head and neck hyperfractionated radiotherapy and / or accelerated
* Head and neck radiotherapy hypofractionated
* Metastatic disease
* Patient deprived of liberty, under guardianship
* Any medical condition or psychological associate that could compromise the patient's ability to participate in the study
* Refusal of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
the proportion of patients with xerostomia | 12 months after completion of radiotherapy.
  Estimate the proportion of patients with xerostomia of grade greater than or equal to 2 assessed by the scale of late toxicity RTOG / EORTC 12 months after completion of radiotherapy.

SECONDARY OUTCOMES:
Evaluation of acute and late xerostomia | after 3, 6 and 12 months after radiotherapy
  Evaluation of acute xerostomia
Measurement of salivary flow with and without stimulation | at 3, 6 and 12 months after end of radiotherapy
  Measurement of salivary flow with and without stimulation
Evaluation of the incidence of acute side effects of radiotherapy | Weekly during radiotherapy
  Evaluation of the incidence of acute and late side effects of radiotherapy
Evaluation of the incidence of late side effects of radiotherapy | At 3, 6 and 12 months after radiotherapy
  Evaluation of the incidence of late side effects of radiotherapy
Evaluation of quality of life and fatigue | At 3, 6 and 12 months after radiotherapy
  Evaluation of quality of life and fatigue
Evaluation of overall survival and progression-free survival | at 3, 6 and 12 months after radiotherapy
  Evaluation of overall survival and progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: bernard GERY, MD, Principal Investigator — Centre François Baclesse
Locations (1):
- Centre François BACLESSE, Caen, France